CLINICAL TRIAL: NCT01287923
Title: Assessment of Biomarkers Initially Identified in Whole Blood by DNA Microarrays in Patients With Aggressive Lymphoma BMS_LyTrans
Brief Title: Assessment of Blood Biomarkers by DNA Microarrays in Patients With Aggressive Lymphoma BMS_LyTrans
Acronym: BMS-LyTrans
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: French Innovative Leukemia Organisation (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010-A00812-37; TRANS/10-01 (Other: Sponsor : Rennes University Hospital); B101038-10 (Other: AFSSAPS References)
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: DLBCL
Keywords: Hematology; Secondary lymphoid organs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For this study, 4 newly included cohorts are necesseray :
  * 100 new DLBCL patients are necessary. The blood will be taken at the diagnosis for DLBCL patients included 075-GOELAMS trial or 075-like patient.
  * 100 healthy blood donors. This cohort of matched for sex & gender will be constituted at the EFS (French Blood Bank) of Rennes.
  * 100 septic patients included at the Rennes University Hospital.
  * 100 075-like DLBCL patients in completed remission.
  This project will also used already available blood collections: 2) Mantle cell lymphoma, 3) localized DLBCL and septic shock. Paraffin blocks of patient 075-trial DLBCLs are in the GOELAMSthèque bank localized in the Pathology Department Hôtel Dieu, Paris supervised by Pr Diane Damotte. Tissue Microarrays and complete paraffin blocks as well as some -80° tumors are already available.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DLBCL: DLBCL patients included 075-GOELAMS trial or 075-like patient.
- Healthy controls: Blood donors from the EFS (French Blood Bank) of Rennes.
- Septic patients: septic patients included at the Rennes University Hospital.
- DLBCL in completed remission: DLBCL patients from the 075 GOELAMS study in completed remission.

SUMMARY:
Diffuse Large B-cell Lymphoma (DLBCL) is the most frequent high grade lymphoma in adults. Although immunotherapy has improved its prognosis, DLBCL is a heterogeneous disease with patients exhibiting a wide range of outcomes with a 5-year overall survival ranging between 55 to 94% depending of the International Prognostic Index factor. Diagnostic and prognostic biomarkers are mandatory to optimize treatment. Transcriptomics has been used to detect such new biomarkers using microarrays analyses applied to RNA collected from total tumor tissues or cell extracts. Molecular prognostic factors have been thoroughly studied in DLBCL tumor tissues. However, it is a big challenge to obtain transcriptomic-qualified tumor samples in a multicentric and prospective clinical trial. Coordinating nvestigator hypothesized that blood may be a deep source of native and secreted analytes and therefore carries transcriptomic signatures related to DLBCL and its prognosis. This project is organized in the extension of the GOELAMS-075 clinical trial which concerns aggressive DLBCL.

DETAILED DESCRIPTION:
Two complementary approaches will be followed, one at the transcriptomic level for confirmation of diagnostic biomarkers and to assess for predictive biomarkers. The other one concern biologic studies to validate our biomarkers at the tissue level. Our project will be organized around 4 workpackages (WP), each of them includes tasks with a specific schedule & predefined deliverables. The first one concerns the general management, data warehouse, collections and different administrative and preanalytic issues. The 3 other WPs are scientific. We are first going to validate a 30-gene list, candidate diagnostic biomarkers, by qRT-PCR on: *) an independent set of DLBCLs compared to matched healthy blood donors (sensitivity assessment) and, **) on a series of low tumor burden DLBCLs, mantle cell lymphomas and non-malignant inflammatory disease constituted by patients with a septic shock (specificity assessment). All this latter collections are already available and ready to use. Secondly, we will complete our series of 89 hybridized patients on AFFY WholeExon microarrays by 60 supplementary and available samples in order to assess for molecular predictor of patient outcome. This question will be address based on the 3-year and 5-year as well, EFS (Event Free Survivor). All the clinical data are available through the GOELAMS eCRF. Since we dispose of a 31 probesets, 30 single genes, signature for the DLBCL diagnosis that involves 9 genes related to the myeloid compartment including 6 genes involved directly or not to the Myeloid-Derived Cell Suppression (MDSC) process, 20 genes described in the context of the cancer and, 11 genes connected to endothelial cells, we decided to explore by flow cytometry blood circulating cells. We will look for myeloid populations & subpopulations, endothelial cells and microparticles. The goal is the identification of specific MDSC perturbations, angiogenic abnormalities and functional impacts on the immune response in the context of the cancer.

We expect by our work to drive both basic science and clinical implications. On the scientific level, blood carries molecular and cellular components involved in tumor-host interactions. Our project should bring a deeper understanding in the immunological response that takes place in the blood compartment. This immunological response will be characterized on a molecular, cellular and functional level. On a clinical point of view, it may bring a new prognostic model in DLBCL. As blood is easily accessible, we expect it to be easily implemented in clinical practice and to allow the design of new clinical trials stratified on tumor biology features. It may also become a new way to monitor DLBCL's response to treatment. Furthermore, this project will provide a large amount of molecular data that can be easily connected with other ongoing GOELAMS studies. Valorisation of our findings will also be serious issue since our project is highly original and valuable.

ELIGIBILITY:
Inclusion Criteria:

* DLBCL or Healthy blood donors or septic patient or GOELAMS 075 patients in completed remission
* Written informed consent

Exclusion Criteria:

* Age < 18 or > 70
* Not written informed consent
* Not affiliated with social security

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DLBCL or Healthy blood donors or septic patient or GOELAMS 075 patients in completed remission
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Research for cancer-related biomarkers | 3 years
  In this project we propose two complementary approaches with a first one orientated to the continuum of our current findings based on genes differentially expressed in blood between DLBCL patients and healthy people and a second one which takes in account the power and originality of our 075 GOELAMS cohort and will be focused on the research of predictive signatures of the DLBCL. We will go beyond the sole transcriptomic approach and also look for relevant cell biology clues.

SECONDARY OUTCOMES:
Sensitivity & specificity of the identified molecular signature in the DLBCL diagnosis context | 3 years
  Sensitivity & specificity of the identified molecular signature in the DLBCL
Identify a prognostic whole blood RNA signature related to aggressive DLBCL | 3 years
  Identify a prognostic whole blood RNA signature related to aggressive DLBCL
Proportion and phenotypic characteristics of circulating cells expressing the previously identified biomarkers at the time of diagnosis of DLBCL | 3 years
  Proportion and phenotypic characteristics of circulating cells expressing the previously identified biomarkers at the time of diagnosis of DLBCL
Immune functions of these circulating cells expressing the previously identified biomarkers at the time of diagnosis of DLBCL | 3 years
  Immune functions of these circulating cells expressing the previously identified biomarkers at the time of diagnosis of DLBCL

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Fest, MD, Principal Investigator — Rennes University Hospital
Locations (17):
- France (17):
  - Amiens University Hospital, Amiens
  - Angers University Hospital, Angers
  - Victor Dupouy Hospital, Argenteuil
  - Cesson-Sévigné Clinic, Cesson-Sévigné
  - La Roche-sur-Yon Hospital, La Roche-sur-Yon
  - Lille University Hospital, Lille
  - Lorient Hospital, Lorient
  - Nantes University Hospital (Hôtel-Dieu), Nantes
  - Bordeaux University Hospital ( Haut-Lévêque Hospital), Pessac
  - Poitiers University Hospital, Poitiers
  - Rennes EFS, Rennes
  - Rennes University Hospital, Rennes
  - Saint-Brieuc Hospital, Saint-Brieuc
  - Loire Cancer Institute, Saint-Priest-en-Jarez
  - Saint-Malo Hospital, St-Malo
  - Toulouse University Hospital, Toulouse
  - Vannes Hospital, Vannes